CLINICAL TRIAL: NCT01331408
Title: An Open, Post-marketing, Multi-center Study to Evaluate Efficacy and Safety of Macrolane VRF30 for Volume Restoration and Contouring of the Buttocks
Brief Title: A Study to Evaluate Efficacy and Safety of Macrolane VRF30 for Volume Restoration and Contouring of the Buttocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 31GC0609
Record Dates: First submitted 2011-04-05; First posted 2011-04-08 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2019-06

CONDITIONS: Volume Restoration and Shaping of the Buttocks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macrolane VRF30 (Experimental): Injection of Macrolane VRF30 in buttocks
  Interventions: Device: Macrolane VRF30

INTERVENTIONS:
Device: Macrolane VRF30 — Injection of Macrolane VRF30 in buttocks. The sum of injected volume of Macrolane VRF30 at initial treatment and touch-up must not exceed 400 ml per Subject

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Macrolane for volume restoration and shaping of the buttocks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years old
* willing to undergo augmentation therapy of the buttocks where a maximum total injected volume of 400 ml of the study product is judged by the Investigator to be enough to achieve full correction
* understand and comply with the requirements of the study
* be willing to understand and comply with the requirements of the study
* be willing to abstain from esthetic surgery and esthetical augmentation procedures (other than the study treatment) between the umbilicus and the knees.
* be a male or non-pregnant, non breast-feeding female.
* give written informed consent to participate in the study

Exclusion Criteria:

* Active skin disease, inflammation or related conditions Tumors or pre-malign tissue disorder near or on the area to be treated
* scar tissue in the area to be treated
* subjects seeking corrections for other body parts then the buttocks anywhere between the umbilicus and the knees
* subjects with human immunodeficiency virus (HIV) associated lipodystrophy
* subjects having undergone liposuction within 6 months prior to inclusion
* BMI <20 or expected instable weight
* insufficient tissue cover in the area to be treated
* excessive skin laxity in the area to be treated
* other injectable implant or permanent implant near or in the area to be treated
* previous radiation therapy of tumors near or in the area to be treated
* concomitant anticoagulant therapy, anti-platelet therapy or a history of bleeding disorders.
* a presence or history of connective tissue diseases
* ongoing immunosuppressive therapy
* known allergies or hypersensitivity reactions towards anesthetics
* previous inflammatory or hypersensitivity reactions towards products containing Hyaluronic acid
* any condition which in the opinion of the investigator makes the subject unsuitable for inclusion use of any investigational drugs or devices within 30 days prior to inclusion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, M.D., Principal Investigator — Akademikliniken, Storängsvägen 10, 115 42 Stockholm, Sweden
Locations (4):
- Artemedis Center for Plastic Surgery, Sint-Denijs-Westrem, Belgium
- Spain (2):
  - Centro Clinico Mir-Mir, Barcelona
  - Cirugia Plastica, Madrid
- Akademikliniken, Stockholm, Sweden

REFERENCES:
- [Result] Camenisch CC, Tengvar M, Heden P. Macrolane for volume restoration and contouring of the buttocks: magnetic resonance imaging study on localization and degradation. Plast Reconstr Surg. 2013 Oct;132(4):522e-529e. doi: 10.1097/PRS.0b013e31829fe47e. PMID 24076699
- [Result] De Meyere B, Mir-Mir S, Penas J, Camenisch CC, Heden P. Stabilized hyaluronic acid gel for volume restoration and contouring of the buttocks: 24-month efficacy and safety. Aesthetic Plast Surg. 2014 Apr;38(2):404-12. doi: 10.1007/s00266-013-0251-9. Epub 2014 Jan 24. PMID 24464121

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Macrolane VRF30
Started | 61
Completed | 50
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Intention To Treat
Arm/Group | Macrolane VRF30
Number analyzed (Participants) | 61
Age, Continuous [Mean (Full Range); unit: years] | 41.3 [20.1 to 64.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement on the Global Esthetic Improvement Scale (GEIS) at Month 6
Description: To evaluate the perceived improvement at 6 months compared to baseline as judged by the Subject using Global Esthetic Improvement Scale (GEIS).
  Percentage of subjects with improved, much improved or very much improved on GEIS, subject's evaluation.
Time Frame: 6 Months
Population: Intention to treat, subjects with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Macrolane VRF30
Number analyzed (Participants) | 56
percentage of participants | 80.4 [67.6 to 89.8]

2. Secondary Outcome: Percentage of Participants With Improvement on the Global Esthetic Improvement Scale (GEIS) at Month 1
Description: To evaluate the perceived improvement at 1 month compared to baseline as judged by the Subject using GEIS.
  Percentage of subjects with improved, much improved or very much improved on GEIS, subject's evaluation.
Time Frame: 1 Month
Population: Intention to treat, subjects with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Macrolane VRF30
Number analyzed (Participants) | 57
percentage of participants | 91.2 [80.7 to 97.1]

3. Secondary Outcome: Percentage of Participants With Improvement on the Global Esthetic Improvement Scale (GEIS) at Month 12
Description: To Evaluate the Perceived Improvement at 12 Months Compared to Baseline as Judged by the Subject Using GEIS.
  Percentage of subjects with Improved, Much Improved or Very Much Improved on GEIS, Subject's evaluation.
Time Frame: 12 Months
Population: Intention To Treat. Subjects with data available
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Macrolane VRF30
Number analyzed (Participants) | 50
percentage of participants | 68.0 [53.3 to 80.5]

ADVERSE EVENTS:
Time Frame: From treatment up to 24 months
Arm/Group | Macrolane VRF30
Serious Adverse Events (participants affected / at risk) | 2/61
Other Adverse Events (participants affected / at risk) | 13/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macrolane VRF30 (N=61)
Lipectomy (Surgical and medical procedures) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macrolane VRF30 (N=61)
Injection Site Pain (General disorders) | 4 (4)
Implant Site Pruritus (General disorders) | 4 (4)
Implant Site Pain (General disorders) | 4 (4)
Implant Site Haematoma (General disorders) | 4 (4)
Implant Site Swelling (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or presentation by PI shall be submitted to Q-Med for review no less than 60 days before submission for publication or presentation. Q-Med will provide any comments to PI within thirty (30) days following receipt of the proposed publication/presentation. PI agree to consider, discuss and give reasonable considerations to comments by Q-Med. Q-Med may also request that the Company name (or that of Q-Med employee) appear or not appear in such publication.